CLINICAL TRIAL: NCT03451799
Title: IIT2016-17-HU-KETORADTMZ: A Phase 1 Study of a 4-month Ketogenic Diet in Combination With Standard-of-care Radiation and Temozolomide for Patients With Newly/Recently Diagnosed Glioblastoma
Brief Title: Ketogenic Diet in Combination With Standard-of-care Radiation and Temozolomide for Patients With Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jethro Hu (Other)
Responsible Party: Sponsor-Investigator, Jethro Hu, Principal Investigator, Faculty, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016-17-HU-KETORADTMZ
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: GBM; Glioblastoma
Keywords: Glioblastoma; Ketogenic diet; Keto diet; GBM
MeSH Terms: conditions — Glioblastoma | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Single arm, prospective cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketogenic diet+radiation+temozolomide (Experimental): Ketogenic diet in combination with standard-of-care radiation and standard-of-care temozolomide
  Interventions: Other: Ketogenic Diet; Radiation: Standard-of-care radiation; Drug: Standard-of-care Temozolomide

INTERVENTIONS:
Other: Ketogenic Diet — A 4-month ketogenic diet will be supervised and monitored by the study investigators. Study dietitians will create personalized meal plans for each patient with the goal of achieving and maintaining metabolic ketosis.
Radiation: Standard-of-care radiation — Patients will receive standard-of-care radiation. Radiation is not protocol directed.
Drug: Standard-of-care Temozolomide — Patients will receive standard-of-care temozolomide. Temozolomide is not protocol directed.

SUMMARY:
Enrolled subjects will be placed on a 16-week ketogenic diet (subject specific as prescribed by RD) while receiving standard of care cancer treatment (Radiation + Temozolomide). Study dietitians will create personalized meal plans for each patient with the goal of achieving and maintaining protocol defined metabolic ketosis. Subjects will be monitored for safety, nutrition, quality of life, and standard of care tumor assessments over the course of the study.

DETAILED DESCRIPTION:
Enrolled subjects will be placed on a 16-week ketogenic diet (subject specific as prescribed by RD) while receiving standard of care cancer treatment (Radiation + Temozolomide). Study dietitians will place patients on a strict and controlled diet that manages daily macronutrient breakdown and increases the ratio of dietary fat relative to protein and carbohydrate consumption. Dietitians will provide guidance and teaching of the diet, as well as, monitoring and diet adjustment to ensure metabolic ketosis. Dietitians and study physicians (and their staff) will monitor subjects for safety, nutrition, quality of life, and standard of care tumor assessments over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Newly or recently diagnosed glioblastoma. Patients may enroll in the study from the time of diagnosis (prior to the initiation of standard-of-care chemoradiation) up until the initiation of post-radiation adjuvant chemotherapy (typically approximately 3-4 weeks after the completion of radiation therapy). Overall, this provides a window of approximately 3 months from the time of diagnosis for patients to enroll in this study. No recurrent glioblastoma is allowed on trial.
* Being seen for treatment of glioblastoma at Cedars-Sinai Medical Center. Note: Okay if patients receiving chemotherapy or radiation therapy at another facility
* Patients on low and managed doses of steroids are permitted. Up to 8 mg dexamethasone or steroid equivalent.

Exclusion Criteria:

* Karnofsky Performance Status of <70 as deemed by physician or equivalent
* Body Mass Index of <22 kg/m2 (rounded to nearest integer)
* Patients with disorders that affect lipid metabolism such as pyruvate carboxylase deficiency, porphyria, primary carnitine deficiency, carnitine palmitoyltransferase I or II deficiency, carnitine translocase deficiency, Beta-Oxidation Defects
* Medical comorbidities that in the opinion of the investigator limits the patient's ability to complete this study
* Pregnant, nursing, or implanted with an intrauterine device (IUD) that is not MR compatible
* Patients who are vegan or vegetarian will be excluded, as the ketogenic diet includes foods that may interfere with these preferences
* Patients on high doses of steroids will be excluded
* Patients currently receiving experimental therapeutic therapy will be excluded from the trial. Note: Off-label therapy use is permitted
* Inability to adhere to the protocol
* Patients with history of allergic reactions to surgical steel or elastomer/rubber are excluded from the activity monitor portion of the study. Because the activity monitor uses a Bluetooth low energy Transceiver, individuals using pacemakers, implantable cardiac defibrillators, neuro-stimulation devices, cochlear implants, hearing aids, or other electronic medical equipment should also be excluded from wearing the activity monitor. They can still use the Aria scale to record weight.
* Patients with mechanically, magnetically, or electrically activated implants, such as cardiac pacemakers, neurostimulators, and infusion pumps, that are not magnetic resonance imaging/positron emission tomography (MRI/PET) compatible.
* Patients with ferromagnetic implants and ferromagnetic foreign bodies, such as intracranial, aneurysm clips, shrapnel and intraocular metal chips as these could become dislodged.
* Patients unable to tolerate MRI/PET imaging secondary to an inability to lie supine or severe claustrophobia as assessed by the treating physician or principal investigator.
* Patients unable to lie still, hold their breath, or follow imaging procedure instructions as assessed by the treating physician or PI.
* Patients whose most recent renal function test does not meet Cedars-Sinai Medical center standard of care MRI contrast protocol requirements (glomerular filtration rate <45ml/min).
* Patients with a known allergy to Fludeoxyglucose F18 (F18-FDG) radioactive tracer or gadolinium-based contrast agent.
* Patients with allergy to animal dander or animal-instigated asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety of the intervention | Four Months
  Proportion of participants experiencing a 10% decrease in weight or body mass index AND have a BMI <18.5 within one month from initiation of the ketogenic diet.
Safety of the intervention | Four months
  Number of related adverse events based on CTCAE v.5.

SECONDARY OUTCOMES:
Feasibility of the intervention | Four Months
  Proportion of enrolled patients able to maintain blood ketone levels >0.3 mM for over 50% of days on study starting 2 weeks after initiation of the ketogenic diet.
Overall Survival | Sixty months
  Time (in months) from initiation of the ketogenic diet to date of death
Time-to-progression | Four Months
  Time (in months) from baseline to progressive disease over study duration (estimated 4 months)
  - measured by RANO criteria (standard of care brain MRI)
Quality of Life (two months) | Two months
  Mean change in overall Quality of Life from baseline to two months.
  -Quality of Life measured using EORTC QLQ-C30 global score
Quality of Life (four months) | Four months
  Mean change in overall Quality of Life from baseline to four months.
  -Quality of Life measured using EORTC QLQ-C30 global score
Cognitive function (Hopkins Verbal Learning Test-Revised) | Four months
  Mean change in cognitive function from initiation of ketogenic diet to four months.
  -measured using Hopkins Verbal learning Test-Revised
Cognitive function (Trail Making Test) | Four months
  Mean change in cognitive function from initiation of ketogenic diet to four months.
  -measured using Trail Making Test
Cognitive function (Controlled Word Association Test) | Four months
  Mean change in cognitive function from initiation of ketogenic diet to four months.
  -measured using Controlled Word Association Test
Cognitive function (Montreal Cognitive Assessment) | Four months
  Mean change in cognitive function from initiation of ketogenic diet to four months.
  -measured using Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jethro Hu, MD, Principal Investigator — Cedars-Sinai Medical Center Samuel Oschin Comprehensive Cancer Institute
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States